CLINICAL TRIAL: NCT01895387
Title: Replacing With Whole Grains and Legumes Reduces Lipoprotein-associated Phospholipase A2 (Lp-PLA2) Activities in Plasma and Peripheral Blood Mononuclear Cells in Patients With Prediabetes or Newly Diagnosed Type 2 Diabetes
Brief Title: Dietary Effects on Circulating Lipoprotein-associated Phospholipase A2 (Lp-PLA2) Activity and Enzyme Activity in Peripheral Blood Mononuclear Cells (PBMCs) in Patients With Prediabetes or Newly Diagnosed Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FN20130614
Record Dates: First submitted 2013-06-14; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Impaired Fasting Glucose; Newly Diagnosed Type 2 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole grains and legumes (Experimental)
  Interventions: Dietary Supplement: Dietary intervention-whole grains and legumes
- Refined rice (Placebo Comparator)
  Interventions: Dietary Supplement: Dietary intervention-Refined rice

INTERVENTIONS:
Dietary Supplement: Dietary intervention-whole grains and legumes — Subjects in the whole-grain group consumed replacing of refined rice intake with 1/3 of legumes, 1/3 of barley, and 1/3 of wild rice three times per day as a carbohydrate source and increased vegetable intake to at least 6 units (30-70 g/unit) per day for sufficient dietary fiber intake.
  Arms: Whole grains and legumes
Dietary Supplement: Dietary intervention-Refined rice — Subjects in the control group maintained their usual diet of refined rice
  Arms: Refined rice

SUMMARY:
We determined the effects of dietary intervention (replacement of refined rice with whole grains and legumes and a high intake of vegetables) on circulating Lp-PLA2 activity and enzyme activity in peripheral blood mononuclear cells (PBMCs) in patients with impaired fasting glucose (IFG), impaired glucose tolerance (IGT) or newly-diagnosed type 2 diabetes.

DETAILED DESCRIPTION:
Ninety-nine patients with impaired fasting glucose (IFG), impaired glucose tolerance (IGT) or newly-diagnosed type 2 diabetes were randomly assigned to either a control group (usual diet with refined rice) or the whole grain group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were in in impaired fasting glucose (IFG, 100≤ fasting glucose <126 mg/dL)
* or newly diagnosed type 2 diabetes (fasting glucose ≥126 mg/dL)

Exclusion Criteria:

* current and/or past history of cardiovascular disease including angina
* liver or kidney dysfunction
* thyroid or pituitary disease
* unstable weight loss/gain (≥2 kg) over the previous 12 months
* pregnancy or lactation
* taking medications or supplements

Ages: 39 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Plasma Lp-PLA2 activity | Change from baseline in Lp-PLA2 at 12 weeks

SECONDARY OUTCOMES:
PBMC Lp-PLA2 activity | Change from baseline in PBMC Lp-PLA2 at 12 weeks

OTHER OUTCOMES:
LDL particle size | Change from baseline in LDL particle size at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph.D, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University, Seoul, South Korea